CLINICAL TRIAL: NCT02316379
Title: Use of Hyperpolarized 129Xe MR Lung Imaging in Adults for Calibration
Acronym: HpXeMRCal
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-7643; IND 123577 (Other: FDA)
Record Dates: First submitted 2014-12-10; First posted 2014-12-12 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2024-04

CONDITIONS: Respiratory Disorders
Keywords: Respiratory
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperpolarized 129 Xenon (Experimental): Administration of up to 1 liter doses of Hyperpolarized Xenon gas during MRI to optimize acquisition of images for adults vs. proton MR imaging. These scans, utilizing volunteers for calibration, may be utilized through this study to optimize the scan details.
  Interventions: Drug: Hyperpolarized 129 Xenon; Device: MRI

INTERVENTIONS:
Drug: Hyperpolarized 129 Xenon — During the scans, subject will inhale hyperpolarized Xenon gas for up to 16 seconds per scan, for up to 4 separate MR scans
  Other Names: HP 129 Xe
Device: MRI

SUMMARY:
The goal of this study is to evaluate the usefulness of hyperpolarized (HP) 129Xe (xenon) gas MRI for regional assessment of lung function in a normal population of adults for the purposes of obtaining optimal images through MRI.

DETAILED DESCRIPTION:
Hyperpolarized 129Xe will be produced, by trained staff, using a polarizer housed at Cincinnati Children's Hospital Medical Center. Individual imaging sessions will be done on a single day and will involve administration of (maximum) 1 liter doses for up to four MRI scans. Subject will inhale hyperpolarized xenon gas and hold breath for up to 16 seconds during the MRI scans. In addition to 129 Xe MRI, a series of anatomical conventional proton MR images may also be collected. Follow up will be done one day and 30 days from the MRI date.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18 years and older
* Participant must be able to hold their breath for up to 16 seconds

Exclusion Criteria:

* History of heart defect
* Pregnancy or positive pregnancy test
* History of uncontrolled asthma defined for this study as requiring use of rescue inhaler ≥ 2 times in past month.
* Symptoms of respiratory infection (loose or productive cough or wheeze), chest tightness, or sinus infection within past week.
* Baseline oximetry at MRI visit of less than 95% on room air or less than 95% on a previously prescribed dosage of oxygen delivered by nasal cannula.
* Participant is claustrophobic and unable to tolerate the imaging.
* Standard MRI exclusions (metal, implants).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-02; Primary Completion 2030-08-24 (Estimated); Study Completion 2031-08-24 (Estimated)

PRIMARY OUTCOMES:
Correlation of ventilated volume predictions obtained with 129Xe MRI vs. 1H MRI | Day 1
  quantify the measurement agreement between the ventilated volume of healthy lungs predicted via 129 Xe MRI and the ventilated volume of the pleural cavity predicted via proton MRI

CONTACTS AND LOCATIONS:
Overall Officials: Jason C Woods, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States